CLINICAL TRIAL: NCT06414499
Title: TNK-tPA Treatment for Acute Minor Ischemic Stroke：A Randomized, Double-blind, Double-dummy Controlled Trial
Brief Title: Teneteplase Reperfusion Therapy in Acute Ischemic Cerebrovascular Events-Ⅳ
Acronym: TRACE Ⅳ
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCRC-2024-03
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Minor Ischemic Stroke
Keywords: minor stroke; tenecteplase
MeSH Terms: interventions — Control Groups; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin combined with clopidogrel (Placebo Comparator): Aspirin 100mg combined with clopidogrel 300mg, plus placebo intravenous rhTNK-tPA
  Interventions: Drug: Control group (Aspirin combined with clopidogrel)
- rhTNK-tPA (0.25 mg/kg) (Experimental): rhTNK-tPA (0.25 mg/kg, max 25 mg) with placebo oral aspirin and clopidogrel
  Interventions: Drug: rhTNK-tPA

INTERVENTIONS:
Drug: rhTNK-tPA — rhTNK-tPA 0.25mg/kg, the maximum dose does not exceed 25mg: 1 vial is dissolved in 3ml of sterile water for injection to prepare a medicinal solution with a concentration of 5.33mg/ml. Calculate the total amount of the drug according to the weight of participant, and the maximum dose shall not exceed 25 mg. It is administered as a single bolus intravenous injection, and the injection is completed within 5-10 seconds. Additionally, placebo oral aspirin and clopidogrel are given. Aspirin 100 mg and clopidogrel 300 mg are administered within 6 ± 2 hours following thrombolytic therapy.
  Arms: rhTNK-tPA (0.25 mg/kg)
Drug: Control group (Aspirin combined with clopidogrel) — Dual antiplatelets with aspirin 100mg and clopidogrel 300mg, plus placebo intravenous rhTNK-tPA. Placebo oral aspirin and clopidogrel are administered within 6 ± 2 hours following intravenous placebo.
  Arms: Aspirin combined with clopidogrel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intravenous tenecteplase (0.25 mg/kg) compared with standard therapy in patients with acute ischemic stroke presenting with mild symptoms-defined as a National Institutes of Health Stroke Scale (NIHSS) score ≤5 accompanied by persistent unilateral limb weakness or speech impairment within 4.5 hours of onset.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized, double-blind, double-dummy controlled (2 arms with 1:1 randomization) trial. Participants with acute minor ischemic stroke (baseline NIHSS≤5) within 4.5 hours of symptoms onset (symptom onset is defined by the "last seen normal" principle for wake-up stroke) will be enrolled. Eligible patients must have neurological deficits involving at least language or motor function. Participants will be randomized into 2 groups: Intervention group (rhTNK-tPA): 0.25mg/kg, the maximum dose does not exceed 25mg, plus placebo oral aspirin and clopidogrel. Aspirin 100mg and clopidogrel 300mg will be given within 6 ± 2 hours after thrombolytic therapy. Control group: Dual antiplatelet therapy with aspirin 100mg and clopidogrel 300mg, plus placebo intravenous rhTNK-tPA. Placebo oral aspirin and clopidogrel will be given within 6 ± 2 hours following the placebo thrombolytic therapy.The primary endpoint is an excellent functional outcome (a modified Rankin Scale score of 0-1) at 90-day.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years;
2. Onset-to-treatment time < 4.5 h; onset time defined as "last known well" time;
3. Clinical diagnosis of minor ischemic stroke (NIHSS ≤ 5) with persistent unilateral limb weakness or speech symptoms, defined as a score of ≥1 on either the language item or a single limb item of the NIHSS;
4. Pre-stroke mRS 0-1;
5. Informed consent signed.

Exclusion Criteria

1. Planned or likely acute endovascular treatments before randomization;
2. NIHSS 1a > 2;
3. Known allergic to rhTNK-tPA;
4. History of intracranial hemorrhage;
5. Severe head trauma or previous stroke within 3 months；
6. Intracranial or spinal surgery within 3 months;
7. Gastrointestinal or urinary tract hemorrhage within 3 weeks；
8. Major surgery within 2 weeks;
9. Arterial puncture at a non-compressible site within 1 week；
10. Intracranial tumors (excluding neuroectodermal tumors, e.g., meningiomas), large intracranial aneurysms, or arteriovenous malformations；
11. Intracranial hemorrhage, including intraparenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, and subdural/epidural hematoma;
12. Active visceral bleeding;
13. Concomitantaortic arch dissection;
14. Acute bleeding tendency, including platelet count <100×10⁹/L or other clinically significant conditions;
15. Uncontrolled hypertension after active antihypertensive treatment: systolic blood pressure >180 mm Hg or diastolic >100 mm Hg;
16. Blood glucose < 2.8 or > 22.2 mmol / L;
17. Prior anticoagulant therapy, such as oral warfarin, with an INR >1.7 or PT >15 seconds;
18. Use of heparin within 24 hours;
19. Use of thrombin inhibitors or factor Xa inhibitors within 48 hours;
20. Large cerebral infarction on head CT or MRI (infarction area >1/3 of the middle cerebral artery territory);
21. Todd's paralysis after a seizure or other neurological/psychiatric disorders affecting cooperation;
22. Severe, uncontrolled infections (e.g., acute pericarditis, infective endocarditis, or acute pancreatitis);
23. Pregnant or breastfeeding women, or women unwilling to use effective contraception during the study period;
24. Participation in another clinical trial within 3 months prior to screening;
25. Other severe illnesses with a life expectancy of less than six months;
26. Deemed unsuitable for the study or at increased risk by the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1386 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Excellent functional outcome (Modified Rankin Scale score, mRS 0-1) at 90-day (± 7 days). | at 90-day (± 7 days)
  Modified Rankin Scale score, mRS 0-1

SECONDARY OUTCOMES:
Good functional outcome (mRS 0-2) at 90-day (± 7 days) | at 90-day (± 7 days)
mRS score at 90-day (± 7 days) | at 90-day (± 7 days)
  shift analysis/ordinal distribution of mRS score at 90-day (±7 days)
COSMOS Scale 0-1 at 90-day (±7days) | 90-day± 7days
COSMOS scale at 90-day (±7 days) | 90-day± 7days
  shift analysis/ordinal distribution of COSMOS scale at 90-day (±7 days)
NIHSS 0-1 at 24-hour, 7-day or before discharge (analyze which occurs first) or/ neurological improvement (NIHSS decreased≥4 from baseline) | at 24-hour, 7-day or before discharge (analyze which occurs first)
Neurological deterioration at 90 days | 90-day (±7 days)
  defined as an increase of ≥4 points in NIHSS score compared to baseline.
New clinical vascular events (ischemic stroke/ hemorrhagic stroke/ myocardial infarction/vascular death) at 90-day (± 7 days), with each vascular event being independently evaluated. | at 90-day (± 7 days)
European quality of life visual analogue scale at 90 days | at 90-day (± 7 days)
Symptomatic intracranial hemorrhage according to the ECASSIII criteria within 36-hour. | within 36-hour
Symptomatic intracranial hemorrhage according to the ECASSIII criteria within 7 days or before discharge. | within 7 days or before discharge
Symptomatic intracranial hemorrhage according to the ECASSIII criteria within 90-day (± 7 days) | within 90-day (± 7 days)
PH2 type intracranial hemorrhage according to the Heidelberg criteria within 90-day (± 7 days) | within 90-day (± 7 days)
Any intracranial hemorrhage within 90-day (± 7 days) | within 90-day (± 7 days)
Severe bleeding events according to the GUSTO criteria within 90-day (± 7 days) | within 90-day (± 7 days)
Total mortality within 90-day (± 7 days) | within 90-day (± 7 days)
Adverse events/Severe adverse events within 90-day (± 7 days) | within 90-day (± 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, PhD, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No